CLINICAL TRIAL: NCT03464825
Title: Prevention of Falls in Older Adults by Specific and Progressive Balance Training
Acronym: BETA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Agneta Stahle, professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K2011-69P-20908-02-4
Record Dates: First submitted 2017-03-03; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Quality of Life

STUDY DESIGN:
Intervention Model Description: One intervention group receiving Specific and progressive balance training One control group
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Participants in the intervention group receive balance training during 3 months 3 times per week
  Interventions: Other: Specific and progressive balance training
- Control (No Intervention): Care as usual

INTERVENTIONS:
Other: Specific and progressive balance training — Specific and progressive balance training for the intervention group
  Arms: Intervention

SUMMARY:
Three months of balance training with follow-up 6 and 12 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* over 60 years with either osteoporosis or Parkinsons disease

Exclusion Criteria:

* under 60 years

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Balance performance - one leg stand | up to 24 months
  One leg stand during 30 seconds

SECONDARY OUTCOMES:
Fear of falling FES-I | up to 24 months
  Questionnaire measuring fear of falling
Health related quality of life - SF-36 | up to 24 months
  Questionnaire measuring health related quality of life

IPD SHARING:
Plan to Share IPD: No